CLINICAL TRIAL: NCT04646759
Title: Fulvestrant or Capecitabine Combined With Pyrotinib in HR-positive and HER2-Positive Metastatic Breast Cancer: A Multicenter, Randomized, Phase III Study
Brief Title: Fulvestrant or Capecitabine Combined With Pyrotinib in HR+/HER2+ Metastatic Breast Cancer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Ying Wang, Associate Professor, Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-KY-140
Record Dates: First submitted 2020-10-27; First posted 2020-11-30 (Actual); Last update posted 2020-11-30 (Actual); Status verified 2020-11

CONDITIONS: Breast Cancer
Keywords: HR-postitive/HER2-positive metastatic breast cancer; fulvestrant; Pyrotinib; capecitabine
MeSH Terms: conditions — Breast Neoplasms | interventions — pyrotinib

STUDY DESIGN:
Intervention Model Description: Patients were randomly assigned to capecitabine plus pyrotinib or fulvestrant plus pyrotinib
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fulvestrant Combined With Pyrotinib (Experimental): Fulvestrant, 500 mg, was injected intramuscularly on D1, D15, D28, D28, once every 28 days； Pyrotinib, 400mg, orally administered daily.
  Interventions: Drug: Fulvestrant combined with Pyrotinib
- Capecitabine Combined With Pyrotinib (Active Comparator): Capecitabine, 1000mg / m^2, twice daily; Pyrotinib, 400mg, orally administered daily.
  Interventions: Drug: Capecitabine combined with Pyrotinib

INTERVENTIONS:
Drug: Fulvestrant combined with Pyrotinib — Fulvestrant 500mg was injected intramuscularly on D1, D15, D28 and D28 Pyrotinib 400mg daily
  Other Names: FASLODEX combined with Pyrotinib
  Arms: Fulvestrant Combined With Pyrotinib
Drug: Capecitabine combined with Pyrotinib — Capecitabine 1000mg/m^2 bid d1-d14，every 21 days Pyrotinib 400mg daily
  Other Names: xeloda combined with Pyrotinib
  Arms: Capecitabine Combined With Pyrotinib

SUMMARY:
Capecitabine combined with pyrotinib is the standard protocol for HR+/HER2+ advanced breast cancer after trastuzumab failure, but the incidence of grade 3 hand-foot-syndrome was 16.4%. Therefore, the search for efficient and low toxicity alternatives has become a research hotspot. Our previous basic studies have shown that ER inhibitor fulvestrant and HER2 inhibitor pyrotinib have a synergistic effect. The preliminary analysis of our prospective shows that the efficacy is close to that of capecitabine combined with pyrotinib, and the adverse events are significantly improved compared with capecitabine combined with pyrotinib. Therefore, it is necessary to further carry out a head-to-head phase III randomized controlled clinical trial to study the efficacy and safety of fulvestrant combined with pyrotinib in the treatment of HR + / HER2 + advanced breast cancer.

DETAILED DESCRIPTION:
Hormone receptor (HR) positive and human epidermal growth factor receptor-2 (HER-2) positive breast cancer has the characteristics of mild biological behavior and slow progression. Currently, capecitabine combined with pyrotinib is the standard protocol for this kind of advanced breast cancer after trastuzumab failure, and the median progression free survival (PFS) is 11.0 months. The incidence of grade 3 hand-foot-syndrome was 16.4%, the incidence of grade 3 diarrhea was 30.6%, and the incidence of grade 3 myelosuppression was 6%. Therefore, the search for efficient and low toxicity alternatives has become a research hotspot.

Our previous basic studies have shown that ER inhibitor fulvestrant and HER2 inhibitor pyrotinib have synergistic effect in inhibiting the proliferation of HR + / HER2 + breast cancer cells. At the same time, the preliminary analysis of our prospective, phase II, single arm study of "Fulvestrant combined with Pyrotinib in the treatment of HR + / HER2 + advanced breast cancer" shows that the efficacy is close to that of capecitabine combined with pyrotinib (median progression free survival is more than 13 months), and the adverse events are significantly improved compared with capecitabine combined with pyrotinib (grade 3 hand-foot-syndrome). This project has been supported by the "Sun-yat sun clinical research and cultivation project" of Sun-Yat Sen Memorial Hospital, Sun-Yat Sen University. Therefore, it is necessary to further carry out a head-to-head phase III randomized controlled clinical trial to study the efficacy and safety of fulvestrant combined with pyrotinib in the treatment of HR + / HER2 + advanced breast cancer, with a non-inferiority cut-off value of HR = 1.30. Combined with the analysis of biomarkers, to find the molecular indicators to predict the benefit of pyrotinib combined with endocrine therapy, so as to provide theoretical basis for guiding precise treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Adult female patients (aged 18-80 years, including 18 and 80 years) with metastatic breast cancer confirmed by pathology or imaging are not suitable for surgical resection or radiotherapy for the purpose of cure;
2. Pathological examination confirmed that ER and / or PR were positive, and HER-2 was positive (ER expression: immunohistochemical staining of tumor cells ≥ 10%; PR expression: immunohistochemical staining of tumor cells ≥ 10%; HER-2 positive: immunohistochemical staining of 3 + or fish positive);
3. Postmenopausal patients (for premenopausal patients, ofs includes bilateral ovariectomy and GnRHa drugs);
4. The disease-free interval between the end of the last trastuzumab and tumor progression was more than 12 months;
5. Trastuzumab has not been treated or only received first-line treatment based on trastuzumab for metastatic diseases, and trastuzumab should be evaluated as effective in the rescue treatment of metastatic breast cancer for the first time.
6. Patients who have received chemotherapy and endocrine therapy in the past (New) adjuvant or for metastatic diseases, and have disease progression during or after treatment;
7. The WHO physical status was 0-2 points, and the expected survival time was not less than 3 months;
8. At least one measurable lesion (short diameter of lymph node ≥ 15mm) was detected in the imaging examination within 2 weeks before enrollment, including normal CT scan ≥ 20 mm, spiral CT scan diameter ≥ 10 mm, or simple bone metastasis.
9. Previous treatment related toxicity should be reduced to NCI CTCAE (version 5.0) ≤ 1 degree (except for hair loss or other toxicity which is judged by the researcher to be safe for the patient)
10. Within one week before admission, blood routine examination was basically normal: A. white blood cell count (WBC) ≥ 3.0 × 10 ^ 9 / L; B. neutrophil count (ANC) ≥ 1.5 × 10 ^ 9 / L; C. platelet count (PLT) ≥ 100 × 10 ^ 9 / L;
11. Liver, kidney and heart function tests were basically normal within one week before enrollment (based on the normal values of laboratories in each research center): A. total bilirubin (TBIL) ≤ 1.5 × upper limit of normal value (ULN), B. alanine aminotransferase (ALT / AST) ≤ 2.5 × ULN (liver metastasis patients ≤ 5xuln), C. serum creatinine ≤ 1.5 × ULN or creatinine clearance rate (CCR) ≥ 60 ml / min; D. left ventricular ejection fraction (LVEF) ≥ 55%, e. QTcF(Fridericia correction) ≤ 470 ms.

Exclusion Criteria:

You cannot be grouped if you meet any of the following:

1. Patients who had not received trastuzumab, chemotherapy and endocrine therapy before;
2. Patients with central nervous system metastasis and clinical symptoms;
3. Patients with visceral crisis;
4. Patients who were considered suitable for chemotherapy by the researchers;
5. There are many factors that affect drug administration and absorption, such as dysphagia, chronic diarrhea and intestinal obstruction.
6. Patients who received radiotherapy, chemotherapy, endocrine therapy, surgery (excluding local puncture) or molecular targeted therapy within 4 weeks before enrollment.
7. He participated in other clinical trials within 4 weeks before enrollment.
8. Patients with metastatic disease received more than first-line endocrine therapy, chemotherapy or targeted therapy.
9. Other malignant tumors in the past 5 years, excluding cured cervical carcinoma in situ, skin basal cell carcinoma or skin squamous cell carcinoma.
10. At the same time, they received any other anti-tumor treatment.
11. Those who have been known to have allergic history to the drug components of this regimen; have a history of immunodeficiency, including HIV positive, HCV, active hepatitis B, or other acquired and congenital immunodeficiency diseases, or have a history of organ transplantation.
12. Severe heart disease or discomfort, including, but not limited to, the following: a history of heart failure or systolic dysfunction (LVEF < 50%); high risk uncontrolled arrhythmias such as atrial tachycardia, resting heart rate > 100bpm, significant ventricular arrhythmias (such as ventricular tachycardia), or higher-level atrioventricular block (i.e., mobitz) The results showed that there was no significant difference between the two groups (systolic blood pressure > 180 mmHg and diastolic blood pressure > 100 mmHg);
13. Pregnant and lactating women, fertile women with positive baseline pregnancy test.
14. According to the judgment of the researchers, there are some accompanying diseases that seriously endanger the safety of patients or affect patients to complete the study.
15. Have a clear history of neurological or mental disorders, including epilepsy or dementia.
16. Any other situation in which the researcher believes that the patient is not suitable for the study, which may interfere with the accompanying diseases or conditions of the study, or have any serious medical obstacles that may affect the safety of the subjects (such as uncontrollable heart disease, hypertension, active or uncontrollable infection, active hepatitis B virus infection)

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 516 (Estimated)
Dates: Start 2020-10-14 (Actual); Primary Completion 2028-12-14 (Estimated); Study Completion 2030-12-14 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | 24 months
  The interval from the date of randomization to the first imaging confirmed progression of disease or death from any cause.
Incidence of grade 3 hand foot syndrome (rate) | From the date of enrollment to one year
  From the date of enrollment to one year, the incidence of grade 3 hand-foot syndrome in the fulvestrant combined with pyrotinib group was compared with that of capecitabine combined with pyrotinib group. The incidence and severity of hand-foot syndrome were evaluated according to CTCAE 5.0 every 9 weeks (± 7 days).

SECONDARY OUTCOMES:
Overall survival (OS) | 50 months
  The time interval from the date of randomization to death due to any cause
Objective response rate (ORR) | 12 months
  According to recist1.1 standard, the proportion of patients whose best remission was CR or PR accounted for the total number of evaluable patients.
Clinical Benefit Rate (CBR) | 12 months
  According to recist1.1 standard, the proportion of patients whose best remission was CR or PR or SD ≥ 24 weeks accounted for the total number of evaluable patients.
Biomarkers and treatment sensitivity analysis | 12 months
  Cox univariate and multivariate analysis will be used to explore the correlation between endocrine and HER2 pathway related biomarkers and treatment sensitivity（The biomarkers to be analyzed included 324 tumor related genes included in the FoundationOne CDx, and ER/PR/HER2/ki67 in IHC）
Quality of life score | 12 months
  Quality of life data will be collected using the following questionnaires: FACT-B score
Incidence of adverse events | from the date of enrollment to one year
  From the date of enrollment to one year, the incidence of adverse events in the fulvestrant combined with pyrotinib group was compared with that of capecitabine combined with pyrotinib group.

CONTACTS AND LOCATIONS:
Overall Officials: Ying Wang, Principal Investigator — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Locations (1):
- Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No
Because the data involves the patient's personal information, it is temporarily decided that we will not disclose the individual participant data.

REFERENCES:
- [Background] Ma F, Ouyang Q, Li W, Jiang Z, Tong Z, Liu Y, Li H, Yu S, Feng J, Wang S, Hu X, Zou J, Zhu X, Xu B. Pyrotinib or Lapatinib Combined With Capecitabine in HER2-Positive Metastatic Breast Cancer With Prior Taxanes, Anthracyclines, and/or Trastuzumab: A Randomized, Phase II Study. J Clin Oncol. 2019 Oct 10;37(29):2610-2619. doi: 10.1200/JCO.19.00108. Epub 2019 Aug 20. PMID 31430226
- [Background] Ma F, Li Q, Chen S, Zhu W, Fan Y, Wang J, Luo Y, Xing P, Lan B, Li M, Yi Z, Cai R, Yuan P, Zhang P, Li Q, Xu B. Phase I Study and Biomarker Analysis of Pyrotinib, a Novel Irreversible Pan-ErbB Receptor Tyrosine Kinase Inhibitor, in Patients With Human Epidermal Growth Factor Receptor 2-Positive Metastatic Breast Cancer. J Clin Oncol. 2017 Sep 20;35(27):3105-3112. doi: 10.1200/JCO.2016.69.6179. Epub 2017 May 12. PMID 28498781
- [Background] Chen Q, Ouyang D, Anwar M, Xie N, Wang S, Fan P, Qian L, Chen G, Zhou E, Guo L, Gu X, Ding B, Yang X, Liu L, Deng C, Xiao Z, Li J, Wang Y, Zeng S, Hu J, Zhou W, Qiu B, Wang Z, Weng J, Liu M, Li Y, Tang T, Wang J, Zhang H, Dai B, Tang W, Wu T, Xiao M, Li X, Liu H, Li L, Yi W, Ouyang Q. Effectiveness and Safety of Pyrotinib, and Association of Biomarker With Progression-Free Survival in Patients With HER2-Positive Metastatic Breast Cancer: A Real-World, Multicentre Analysis. Front Oncol. 2020 May 25;10:811. doi: 10.3389/fonc.2020.00811. eCollection 2020. PMID 32528890
- [Background] Lin Y, Lin M, Zhang J, Wang B, Tao Z, Du Y, Zhang S, Cao J, Wang L, Hu X. Real-World Data of Pyrotinib-Based Therapy in Metastatic HER2-Positive Breast Cancer: Promising Efficacy in Lapatinib-Treated Patients and in Brain Metastasis. Cancer Res Treat. 2020 Oct;52(4):1059-1066. doi: 10.4143/crt.2019.633. Epub 2020 Apr 24. PMID 32340083
- [Background] Johnston SRD, Hegg R, Im SA, Park IH, Burdaeva O, Kurteva G, Press MF, Tjulandin S, Iwata H, Simon SD, Kenny S, Sarp S, Izquierdo MA, Williams LS, Gradishar WJ. Phase III, Randomized Study of Dual Human Epidermal Growth Factor Receptor 2 (HER2) Blockade With Lapatinib Plus Trastuzumab in Combination With an Aromatase Inhibitor in Postmenopausal Women With HER2-Positive, Hormone Receptor-Positive Metastatic Breast Cancer: ALTERNATIVE. J Clin Oncol. 2018 Mar 10;36(8):741-748. doi: 10.1200/JCO.2017.74.7824. Epub 2017 Dec 15. PMID 29244528 (Retraction: PMID 32822279 J Clin Oncol. 2021 Jan 1;39(1):95)
- [Background] Robertson JFR, Steger GG, Neven P, Barni S, Gieseking F, Nole F, Pritchard KI, O'Malley FP, Simon SD, Kaufman B, Petruzelka L. Activity of fulvestrant in HER2-overexpressing advanced breast cancer. Ann Oncol. 2010 Jun;21(6):1246-1253. doi: 10.1093/annonc/mdp447. Epub 2009 Oct 29. PMID 19875750
- [Background] Tolaney SM, Wardley AM, Zambelli S, Hilton JF, Troso-Sandoval TA, Ricci F, Im SA, Kim SB, Johnston SR, Chan A, Goel S, Catron K, Chapman SC, Price GL, Yang Z, Gainford MC, Andre F. Abemaciclib plus trastuzumab with or without fulvestrant versus trastuzumab plus standard-of-care chemotherapy in women with hormone receptor-positive, HER2-positive advanced breast cancer (monarcHER): a randomised, open-label, phase 2 trial. Lancet Oncol. 2020 Jun;21(6):763-775. doi: 10.1016/S1470-2045(20)30112-1. Epub 2020 Apr 27. PMID 32353342